CLINICAL TRIAL: NCT05169476
Title: Potential Fall Risk Increasing Drugs and Falls in Community-dwelling Older Adults: A Prospective Cohort Study
Brief Title: FRIDs and Fall Risk Among Older Adults
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Gustav Valentin Blichfeldt Sørensen, MD, PhD, Aalborg University Hospital
Other Study IDs: 20155750
Record Dates: First submitted 2021-12-10; First posted 2021-12-27 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Fall; Fall Injury; Aging; Aged; Medication
Keywords: Older adults; Accidental falls; Fall-risk increasing drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The European Geriatric Medicine Society (EuGMS) Task and Finish Group published a consensus paper on fall-risk increasing drugs. However, the group did not reach consensus on 17 medication classes as potential FRIDs. Thus, in this study the investigators want to examine the association between use of these potential FRIDs and falls rate with a 1-year follow-up in a cohort of community-dwelling older adults, aged 75 years or more.

DETAILED DESCRIPTION:
Falls in community-dwelling older adults are the most frequent cause of injury. Every year, 30% of the adults over the age of 65 years fall increasing to 32-42% among those aged ≥ 75 years. Most falls have a multifactorial aetiology such as previous falls, advanced age, cognitive impair-ment, environmental risks, and hazardous activities, along with presence of chronic disease, muscle weakness, gait and balance disorders, and medication use Especially the use of fall-risk-increasing drugs (FRIDs) is a prominent risk factor.

Recently, The European Geriatric Medicine Society (EuGMS) Task and Finish Group published a consensus paper classifying 14 medication classes as fall-risk-increasing drug (FRID) (14). Most of them were psychotropics, but several new possible FRIDs were identified. However, the group did not reach consensus on 17 medication classes as potential FRIDs.

Therefore, to achieve a better understanding of these 17 medication classes as potential FRIDs, more studies taking these issues into account are warranted.

Primary objective:

To examine the association between use of the potential FRIDs and falls rate with a 1-year follow-up in a cohort of community-dwelling older adults, aged 75 years or more.

Study design and sample:

A prospective cohort study with 1-year follow-up will be performed in collaboration with the municipality of Hjørring, Denmark. The sample size was derived without a recommended power calculation; hence, the sample size builds on feasible recruitment within the 13 months inclusion period granted by the municipality due to economical and administrative reasons.

Study setting, participants, data collectors, process of recruitment and data collection:

According to Danish legislation on health and social services, Danish municipalities are responsible for developing and initiating prophylactic and health-promoting initiatives for their senior citizens. This is done through different authorities in the municipality (e.g. preventive-home-visits, senior activity centres). Also, the municipality of Hjørring administers a local hall for citizens together with general- and patient associations. Therefore, data collection will be performed in participants' own homes through preventive-home-visits, at senior activity centres and at the local hall in the municipality of Hjørring, Denmark.

Baseline characteristics:

Data collection was performed at baseline and based on a multifactorial falls risk test battery in-cluding various physical tests (static balance under dual-task conditions, grip- and lower limb strength, reaction time of lower limbs and gait speed); self-report questionnaire on sociodemo-graphic characteristics, frailty, nutrition, disability, fear of falling, health-related quality of life, depressive symptoms, several physical symptoms, cognitive tests; and reporting of comorbidities (23). The participants' comorbidities were obtained from the participants' hospital records and the diagnoses were indexed according to the International Classification of Diseases 10th revision (ICD-10).

Baseline medication:

To determine the participants' medications at inclusion, the investigators consulted the national Shared Medica-tion Record (SMR). The SMR is a national registry of current medication use and pharmacy rec-ords of prescriptions to each citizen in Denmark. Any physician involved in the patients' clinical course has access to the SMR data and all details of each prescription and the date of the latest medication reconciliation are provided (24). For each participant all medication registered in SMR at baseline was documented and indexed according to the WHO-recommended anatomical therapeutic chemical (ATC) medication classification system.

Confounding covariates:

Many different risk factors and predictors for falls in older adults have been described previously. All these risk factors are possible confounders to the potential FRIDS; hence, the following a priori list specifies the confounding variables to be adjusted for in the multivariate regression model:

* Age
* Sex
* History of previous falls
* The comorbidity related to the potential FRID to adjust for confounding by indication
* Fear of falling using Short Falls Efficacy Scale-International 7-item
* Gait speed measured with a 4-meter walk test
* Cognitive impairment estimated by the Orientation-Memory-Concentration test per-formed over the telephone
* Frailty using the Tilburg Frailty Indicator
* Physical and instrumental disability in activities of daily living using the Vulnerable El-ders Survey 13 .
* Depressive symptoms using Geriatric Depression Scale 4 item, a depression diagnosis or prescription of any antidepressants
* Use of benzodiazepines, benzodiazepines derivatives or non-benzodiazepines (Z-drugs)
* Use of opioids

ELIGIBILITY:
Inclusion criteria:

* Community-dwelling older adults
* 75 years old or above

Exclusion criteria:

* Presence of acute illness defined by the presence of a participant-reported experience of illness arisen within 7 days prior to inclusion impairing their everyday functioning in such a way that they opt out of social activities outside their homes while this state is present.
* Unable to understand Danish evaluated by the data collectors.
* Diagnosed with dementia.
* Unable to stand up for 60 seconds without support and visually fixate on an object at the same time. Support is defined by any assistive devices or help from another person.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The target group of PHVs is community-dwelling older adults primarily +75 years old. PHVs are not offered to citizens already receiving local authority home help except for those receiving help with cleaning. As of 2017, the target group of PHVs in the municipality of Hjørring consisted of approximately 4,800 community-dwelling older adults of which 2,053 received a PHV.
  The target group of SACs is primarily retirees (+65 years old), but also early retirees (+60 years old) with reduced physical, psychological or social functional capacity. As of 2018, 318 citizens of the target group attend SACs in the municipality of Hjørring weekly.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-07-18 (Actual); Study Completion 2020-07-18 (Actual)

PRIMARY OUTCOMES:
Number of falls | 1-year follow-up
  Falls will be monitored using monthly prepaid fall calendars and validated by a phone call if a fall is registered. Also, circumstances of the fall will be asked about in the phone call.
  Blinding:
  Assessors of the outcome will be naturally blinded towards the predictors due to test results not being available before end of follow-up. Also, assessors of the outcome will be blinded to the questionnaire results by not having access to these in REDCap

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Aktivitetscenter Lynggården, Hirtshals
  - Aktivitetscenter Vesterlund, Hjørring
  - Forsamlingsbygningen, Hjørring
  - Sundhedscenter Hjørring, Hjørring
  - Sindal aktivitetscenter, Sindal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT05169476/Prot_SAP_001.pdf